CLINICAL TRIAL: NCT05867888
Title: Effect of Shock Wave Therapy Versus Low Level Laser Therapy in Patients With Plantar Fasciitis
Brief Title: Shock Wave Therapy Versus Low Level Laser Therapy in Patients With Plantar Fasciitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reham Mohamed Lotfy Soliman, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004154
Record Dates: First submitted 2023-04-29; First posted 2023-05-22 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Plantar Fascitis
Keywords: low level laser therapy; shock wave therapy; stretching exercises
MeSH Terms: interventions — Extracorporeal Shockwave Therapy; Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): conventional physical therapy program (Instructions, Ice application, Deep tissue massage, Stretching exercises, Joint mobilization and isometric exercises).
  Interventions: Other: conventional therapy
- Experimental group 1 (Experimental): Shock wave therapy + Conventional physical therapy.
  Interventions: Other: conventional therapy; Other: shock wave therapy
- Experimental group 2 (Experimental): Low level laser therapy + Conventional physical therapy.
  Interventions: Other: conventional therapy; Other: low level laser therapy

INTERVENTIONS:
Other: conventional therapy — conventional therapy ( instructions, ice application, deep tissue massage, stretching exercises, joint mobilization and isometric exercises )
Other: shock wave therapy — Acoustic waves (shock waves) that can carry energy and can propagate through tissues promote healing effects.
  Arms: Experimental group 1
Other: low level laser therapy — The application of light to a biologic system to promote tissue regeneration, reduce inflammation and relieve pain.
  Arms: Experimental group 2

SUMMARY:
Both shock wave therapy and low level laser therapy in plantar fasciitis are effective in improvement of such cases without any side effects but there are no previously published studies on the use of shock wave therapy versus low level laser therapy in plantar fasciitis and, hence, evidence of its acceptability and effectiveness compared with each other remains to be established.

DETAILED DESCRIPTION:
Plantar fasciitis is a result of degenerative irritation of the plantar fascia origin at the medial calcaneal tuberosity of the heel as well as the surrounding perifascial structures, it is a common problem accounting for approximately one million patient visits per year, it is often an overuse injury. As a result tight gastrocnemius, soleus, and/or other posterior leg muscles have also been commonly found in patients with this condition.

Shock wave therapy is thought to provide long lasting analgesia and stimulate the healing process, Low level laser therapy has been used to relieve pain caused by plantar fasciitis, also stretching of the shortened and contracted plantar flexors may positively influence an individual's functional activities of daily living and decrease the risk of injury.

ELIGIBILITY:
Inclusion Criteria:

1. Age ranges from 40-60 years old.
2. Both genders will be included.
3. Unilateral plantar fasciitis.
4. Duration of symptoms more than 4 weeks.
5. Positive Windlass test and negative Tinel and calcaneus squeeze tests.
6. Patients will be classified according to their BMI (18.5 - 24.9) kg/m2

Exclusion Criteria:

1. Open wound, infection in plantar surface of foot.
2. History of foot surgery.
3. History of trauma or fracture in foot or ankle.
4. Neuropathic pain as diabetes mellitus.
5. Peripheral vascular disease.
6. Calcaneal stress fracture or show evidence of a foreign body or tumor of the affected heel.
7. Previously suffered a rupture or surgery of the plantar fascia. Existing or prior osteomyelitis of the involved calcaneus.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Assess the change in pain intensity level | Before treatment and after 6 weeks treatment
  The visual analogue scale (VAS) is a widely utilized pain intensity level assessment instrument in patients with plantar fasciitis. The visual analogue scale (VAS) is typically composed of a horizontal line from zero (minimum value) to 10 (maximum value) where zero signifies (no pain) and 10 signifies (worst pain) one can imagine.
Assess the change in pain pressure threshold | Before treatment and after 6 weeks treatment
  Pressure algometry will be used to evaluate the pain pressure threshold for the two predetermined locations on the affected leg: gastrocnemius (middle point over the muscle belly) and soleus (center point of the muscle belly 10 cm above the Achilles tendon). The participant will speak up at the point where the pressure evoke a painful sensation. This process will be repeated 3 times in the same manner, and three measurements will be recorded at the same point on the plantar fascia. An average of the three readings will be recorded. Higher algometer scores indicate greater pressure threshold, therefore less tenderness. Lower algometer scores indicate less pressure threshold, thus more tenderness.
Assess the change in range of ankle motion | Before treatment and after 6 weeks treatment
  Ankle range of motion (ROM) will be measured by using digital goniometer (ankle dorsiflexion and plantarflexion ranges will be measured). It can monitor the progress of intervention.
Assess the change in foot functional disability | Before treatment and after 6 weeks treatment
  Foot functional disability will be assessed by foot and ankle ability measure questionnaire (FAAM). Higher scores on the questionnaire indicate a higher level of physical functioning and lower scores on the questionnaire indicate a lower level of physical functioning.
Assess the change in ankle stability | Before treatment and after 6 weeks treatment
  The Human Assessment Computer (HUMAC) Balance System will be used in the current study to assess limits of stability of ankle joint.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma S Amin, Professor, Study Chair — Cairo University; Rania N Karkousha, Ass.prof, Study Director — Cairo University; Mohamed I Abd Elhay, Lecturer, Study Director — Cairo University; Ashraf N Moharram, Professor, Study Director — Cairo University
Locations (1):
- Reham, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No